CLINICAL TRIAL: NCT02669407
Title: Splanchnic Nerve Block for Acute Heart Failure
Brief Title: Splanchnic Nerve Anesthesia in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00066528
Record Dates: First submitted 2016-01-22; First posted 2016-02-01 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regional nerve anesthesia (Experimental): Regional nerve anesthesia of splanchnic nerve
  Interventions: Procedure: splanchnic nerve anesthesia with a local anesthetic; Drug: regional nerve block with a local anesthetic (Lidocaine)

INTERVENTIONS:
Procedure: splanchnic nerve anesthesia with a local anesthetic — regional nerve block of the splanchnic nerve
Drug: regional nerve block with a local anesthetic (Lidocaine)

SUMMARY:
Patients admitted for acute heart failure and undergoing right heart catheterization will be enrolled in this study. Subjects will undergo catheterization of the heart to obtain central cardiac pressure and other cardiac hemodynamic parameters. Subsequently, the subject will undergo a regional nerve block of the splanchnic nerves. Patients will remain in the catheterization lab for the duration of anesthetic block and will be continuously hemodynamically monitored.

This study will be a prospective, uncontrolled clinical trial. The study will not be controlled as invasive monitoring of hemodynamics will be performed, allowing clear demonstration of a cause-effect relationship. The goal of the study is to provide proof of concept.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure (HF)
* Prior admissions for decompensated HF
* Symptomatic with dyspnea with clinical, radiographic or echocardiographic signs of fluid overload
* On a stable HF drug regimen prior to admission
* Anticipated hospital stay of at least 2 nights following catheterization procedure

Exclusion Criteria:

* Ongoing treatment with oral anticoagulation other than aspirin
* Immunosuppressive medications for solid organ transplant
* Acute MI (STEMI or NSTEMI) within 7 days
* Evidence of cardiogenic shock within 48 hours
* Systolic blood pressure < 90 mmHg or >180 mmHg
* Restrictive or constrictive cardiomyopathy
* Chronic kidney disease stage 3 or higher due to primary renal pathology
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01-01; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke, Durham, North Carolina, United States

REFERENCES:
- [Derived] Fudim M, Patel MR, Boortz-Marx R, Borlaug BA, DeVore AD, Ganesh A, Green CL, Lopes RD, Mentz RJ, Patel CB, Rogers JG, Felker GM, Hernandez AF, Sunagawa K, Burkhoff D. Splanchnic Nerve Block Mediated Changes in Stressed Blood Volume in Heart Failure. JACC Heart Fail. 2021 Apr;9(4):293-300. doi: 10.1016/j.jchf.2020.12.006. Epub 2021 Mar 10. PMID 33714749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited patients hospitalized for acute decompensated heart failure (ADHF) at Duke University Hospital between April 2017 and May 2018.
Groups:
- Regional Nerve Anesthesia: Regional nerve anesthesia of splanchnic nerve
  splanchnic nerve anesthesia with a local anesthetic: regional nerve block of the splanchnic nerve
  regional nerve block with a local anesthetic (Lidocaine)
Period: Overall Study
Arm/Group | Regional Nerve Anesthesia
Started | 14
Completed | 11
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Central Venous Pressure [Mean (Standard Deviation); unit: mmHg] | 18.73 (5.57)
Pulmonary Arterial Mean Pressure [Mean (Standard Deviation); unit: mmHg] | 45.45 (5.99)
Pulmonary Capillary Wedge Pressure [Mean (Standard Deviation); unit: mmHg] | 30 (7)

OUTCOME MEASURES:

1. Primary Outcome: Central Venous Pressure
Time Frame: Baseline, 90 minutes
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
mmHg
  Baseline | 18.73 (5.57)
  90 minutes | 14.91 (5.24)

2. Primary Outcome: Pulmonary Arterial Mean Pressure
Time Frame: baseline, 30 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
mmHg
  Baseline | 45.45 (5.99)
  30 minutes | 37.64 (7.03)
Statistical Analysis 1: Comparison: Regional Nerve Anesthesia; Test type: Other — Single group; p < 0.001, Tukey's method

3. Primary Outcome: Pulmonary Capillary Wedge Pressure
Time Frame: baseline, 30 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
mmHg
  Baseline | 30 (7)
  30 minutes | 22 (7)
Statistical Analysis 1: Comparison: Regional Nerve Anesthesia; Baseline, 30 minutes; Test type: Other — Single group; p = 0.001, Tukey's method

4. Secondary Outcome: Cardiac Index
Time Frame: baseline, 30 minutes
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
L/min/m^2
  Baseline | 2.17 (0.74)
  30 minutes | 2.59 (0.65)
Statistical Analysis 1: Comparison: Regional Nerve Anesthesia; baseline, 30 minutes; Test type: Other — Single group; p = 0.007, Tukey's method

5. Secondary Outcome: Ejection Fraction (LVEF)
Time Frame: Baseline, 90 minutes
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: percentage of ejected blood per contract
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
percentage of ejected blood per contract
  Baseline | 18.27 (11.18)
  90 minutes | 19.4 (10.32)

6. Secondary Outcome: Pulmonary Artery Systolic Pressure
Time Frame: Baseline, 30 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
mmHg
  Baseline | 65.18 (9.95)
  30 minutes | 53.91 (12.47)

7. Secondary Outcome: Right Ventricular Diameter
Time Frame: Baseline, 30 mins
Population: Data not collected
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 0

8. Secondary Outcome: Left Ventricular Diameter
Time Frame: Baseline, 30 mins
Population: Participants who completed the study
Measure: Median (Standard Deviation); unit: cm
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
cm
  Left ventricular end diastolic dimension; Baseline | 6.2 (1.0)
  Left ventricular end diastolic dimension; 30 mins | 6.1 (0.9)
  Left ventricular end systolic dimension; Baseline | 5.4 (1.3)
  Left ventricular end systolic dimension; 30 mins | 5.4 (1.3)
Statistical Analysis 1: Comparison: Regional Nerve Anesthesia; Change in left ventricular end diastolic dimension; Test type: Other — Single group; p = 0.237, t-test, 2 sided
Statistical Analysis 2: Comparison: Regional Nerve Anesthesia; Change in left ventricular end systolic dimension; Test type: Other — Single group; p = 0.586, t-test, 2 sided

9. Secondary Outcome: N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) Level
Description: NT-proBNP level is elevated in heart failure and reflects its severity. A higher value indicates less stability.
Time Frame: Baseline; 90 minutes
Population: Participants who completed the study.
Measure: Median (Inter-Quartile Range); unit: pg/dL
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
pg/dL
  Baseline | 4,297 [1,656 to 10,842]
  90 minutes | 2,936 [1,317 to 7,136]
Statistical Analysis 1: Comparison: Regional Nerve Anesthesia; Test type: Other — Single group; p = 0.175, t-test, 2 sided

10. Secondary Outcome: Urine Output Measured in ml Over 3 Hours
Time Frame: Baseline, post-procedure (0-3 hours)
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: ml over 3 hours
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
ml over 3 hours
  Baseline | 138.09 (92.22)
  post-procedure 0-3 hours | 258.64 (199.22)

11. Secondary Outcome: Change in Blood Urea Nitrogen (BUN)
Description: BUN represents the major nitrogen excretion pathway and is used to evaluate renal function. Higher BUN levels indicate less stability.
Time Frame: Baseline; 90 minutes
Population: Participants who completed the study.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
mg/dL
  Baseline | 61 [31 to 68]
  90 minutes | 53 [26 to 68]
Statistical Analysis 1: Comparison: Regional Nerve Anesthesia; Test type: Other — Single group; p = 0.061, t-test, 2 sided

12. Secondary Outcome: Change in Creatinine Level
Description: Creatinine measurements are used to evaluate renal function. Higher creatinine levels indicate less stability.
Time Frame: Baseline; 90 minutes
Population: Participants who completed the study.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
mg/dL
  Baseline | 2.1 [1.5 to 2.6]
  90 minutes | 1.9 [1.4 to 2.7]
Statistical Analysis 1: Comparison: Regional Nerve Anesthesia; Test type: Other — Single group; p = 0.787, t-test, 2 sided

13. Secondary Outcome: Dyspnea as Measured on Likert Scale
Description: The scale ranges from -3 (markedly worse) to 3 (markedly improved). 0 = no change.
Time Frame: 15, 30, 45, 60, 75, 90 minutes; 24 hours
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
Participants
  15 minutes: 3=Markedly improved | 2
  15 minutes: 2=Moderately Improved | 1
  15 minutes: 1=Minimally improved | 4
  15 minutes: 0=No change | 4
  15 minutes: -1=Minimally worse | 0
  15 minutes: -2=Moderately worse | 0
  15 minutes: -3=Markedly worse | 0
  30 minutes: 3=Markedly improved | 0
  30 minutes: 2=Moderately Improved | 3
  30 minutes: 1=Minimally improved | 5
  30 minutes: 0=No change | 2
  30 minutes: -1=Minimally worse | 1
  30 minutes: -2=Moderately worse | 0
  30 minutes: -3=Markedly worse | 0
  45 minutes: 3=Markedly improved | 0
  45 minutes: 2=Moderately Improved | 3
  45 minutes: 1=Minimally improved | 7
  45 minutes: 0=No change | 1
  45 minutes: -1=Minimally worse | 0
  45 minutes: -2=Moderately worse | 0
  45 minutes: -3=Markedly worse | 0
  60 minutes: 3=Markedly improved | 0
  60 minutes: 2=Moderately Improved | 1
  60 minutes: 1=Minimally improved | 5
  60 minutes: 0=No change | 4
  60 minutes: -1=Minimally worse | 1
  60 minutes: -2=Moderately worse | 0
  60 minutes: -3=Markedly worse | 0
  75 minutes: 3=Markedly improved | 1
  75 minutes: 2=Moderately Improved | 2
  75 minutes: 1=Minimally improved | 3
  75 minutes: 0=No change | 5
  75 minutes: -1=Minimally worse | 0
  75 minutes: -2=Moderately worse | 0
  75 minutes: -3=Markedly worse | 0
  90 minutes: 3=Markedly improved | 3
  90 minutes: 2=Moderately Improved | 2
  90 minutes: 1=Minimally improved | 3
  90 minutes: 0=No change | 3
  90 minutes: -1=Minimally worse | 0
  90 minutes: -2=Moderately worse | 0
  90 minutes: -3=Markedly worse | 0
  24 hours: 3=Markedly improved | 3
  24 hours: 2=Moderately Improved | 2
  24 hours: 1=Minimally improved | 5
  24 hours: 0=No change | 0
  24 hours: -1=Minimally worse | 0
  24 hours: -2=Moderately worse | 0
  24 hours: -3=Markedly worse | 1

14. Secondary Outcome: Change in Clinical Symptoms, as Measured by 6 Minute Walk Test
Description: The 6 Minute Walk Test (6MWT) is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Time Frame: Baseline, 90 minutes, 24 hours
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Regional Nerve Anesthesia
Number analyzed (Participants) | 11
meters
  Baseline, 90 minutes | 8.7 (51.6)
  Baseline, 24 hours | 24.7 (31.2)
Statistical Analysis 1: Comparison: Regional Nerve Anesthesia; Baseline, 90 minutes; Test type: Other — Single group; p = 0.606, t-test, 2 sided
Statistical Analysis 2: Comparison: Regional Nerve Anesthesia; Baseline, 24 hours; Test type: Other — Single group; p = 0.045, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Regional Nerve Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT02669407/Prot_SAP_000.pdf